CLINICAL TRIAL: NCT06005506
Title: 'sPATIALS3' - National Multicenter Randomized Controlled Interventional Study, Comparing an Active Symbiotic and a Passive Symbiotic Aimed at Evaluating the Effect on the Intestinal Microbiota and on the State of Health and Well-being of Various Types of Chronically Frail Patients United by Alterations of Intestinal Function.
Brief Title: National Multicenter Interventional Study Aimed at Evaluating the Effect on the Intestinal Microbiota in Chronically Frail Patients Who Share Alterations in Intestinal Function.
Acronym: sPATIALS3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Biomedical Technologies-National Research Council, Italy (Other)
Collaborators: Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other); IRCCS Eugenio Medea (Other); Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NM102_SPATIALS3
Record Dates: First submitted 2023-07-10; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Adhd; ALS; Bronchial Asthma
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Asthma | interventions — Dietary Fiber; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic + fiber (Active Comparator): These subjects will be given a passive symbiotic preparation again consisting of two sticks of 1500mg each to be taken once a day:
  * Purple Sachet - Prebiotic - Composed of 500mg acacia fiber (Fibregum®) with high prebiotic activity and 500mg mai starch. Excipients and flavorings.
  * White Sachet - Probiotic - 30 Billion bacterial strains Lactobacillus plantarum LP (PBS067- EU Collection DSM 24937), Lactobacillus acidophilus L.
  Interventions: Dietary Supplement: Dietary fiber; Dietary Supplement: Probiotic
- Probiotic + Prebiotic (Experimental): These subjects will be given an active symbiotic preparation consisting of two differently colored sticks of 1500mg each to be taken once a day:
  * Purple Sachet - Active Prebiotic - 500 mg of Fibregum®, a slow-fermenting prebiotic fiber and 500 mg of standardized extract of pigmented Zea Mays L fruit, rich in anthocyanins and polyphenols. Excipients and flavorings.
  * White Sachet - Probiotic - 30 Billion Bacterial Strains Lactobacillus plantarum LP (PBS067- EU Collection DSM 24937), Lactobacillus acidophilus LA (PBS066 - EU Collection DSM 24936) and Bifidobacterium animalis subsp. lactis BL (BL050 - Eu Collection DSM 25566).
  Interventions: Dietary Supplement: Prebiotic fiber; Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic fiber — Moradyn active prebiotic fiber product
  Arms: Probiotic + Prebiotic
Dietary Supplement: Dietary fiber — Fibregum non-active fiber product
  Arms: Probiotic + fiber
Dietary Supplement: Probiotic — Defense Plus probiotic complex

SUMMARY:
The objective of the study will be to understand whether a supplementation of the diet with an active symbiotic, i.e. characterized by a mix of probiotics and a specially selected fiber with prebiotic activity combined with a vegetable extract with beneficial activities on carbohydrate and lipid metabolism, can reduce the relative inflammatory potential and improve absorption, intestinal motility and bowel habit of patients with various pathological conditions, such as ALS, ADHD and bronchial asthma.

DETAILED DESCRIPTION:
Clinical survey conducted for research and study purposes, multicenter, focusing on ALS patients, elderly patients with chronic diseases, and pediatric patients with neurodevelopmental disorders. For each of the diseases treated, patients will be randomized into the two treatment arms (Study Group, GS; Control Group, GC) according to a block randomization, with a block size of 4 and an allocation ratio of 1:1. The randomization will be double-blind.

* Study Group or GS: These subjects will be given an active symbiotic preparation consisting of two sticks of 1500mg each and of different colors.
* Control group or GC:These subjects will be given a passive symbiotic preparation again consisting of two sticks of 1500mg each.

ELIGIBILITY:
Population 1 : ALS

Inclusion Criteria:

* Age at enrollment ≥18 years;
* ALS diagnosis defined or probable according to El Escorial criteria (Brooks et al., 2000);
* Respiratory function with FVC% >50%.

Exclusion Criteria:

* Subjects unable to give informed consent to the study;
* presence of psychiatric disease or severe cognitive impairment;
* presence of tracheotomy; presence of severe pre-existing gastrointestinal disease (e.g., ulcerative rectocolitis; Crohn's disease).

Population 2: ADHD

Inclusion Criteria:

* children between 6 and 16 years old
* children with ADHD, diagnosed with DSM-5 criteria and in accordance with the protocol shared by the Regional ADHD Reference Centers Lombardy.

Exclusion Criteria:

* presence of intellectual disability (QIT<70),
* presence of neurological diseases, epilepsy
* presence of genetic syndromes
* treatment with drug therapies.

Co-diagnosis with other psychiatric or neurodevelopmental disorders (i.e. Autism, Anxiety, Depression etc) will not be considered a criterion of exclusion.

Population 3: Bronchial Ashtma

Inclusion Criteria:

* adults above 18 years of age
* diagnosed with Bronchial Ashtma following ERS-ETS criteria

Exclusion Criteria:

* life expectancy less than 18 months
* active respiratory infections
* cognitive disorders that prevent participation to the study (MMS <24)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in levels of Short Chain Fatty Acids (SCFA) | Before and After 3 months of intervention
  Evaluation of pre-post treatment variation of the level of specific SCFAs (acetic acid, propionic acid, butyric acid and valeric acid) both within the group of the treated and between the group of treated patients and the placebo group.
Change in levels of branched chain fatty acids (isobutyrate and isovalerate) | Before and After 3 months of intervention
  Evaluation of the pre-post nutritional variation of the level of branched chain fatty acids (isobutyrate and isovalerate) between the group of treated patients and the placebo group

SECONDARY OUTCOMES:
Conners' Parent Rating Scale-Revised - scale H (ADHD Index) | Before and After 3 months of intervention
  The score of subscale H on the Conners' Parent Rating Scale-Revised allows to identify children / adolescents at risk of ADHD.
  The score is a T-score with mean 50 and deviation standard 10 in the general population Minimum score = 35 Maximum score = 100
  Higher scores correspond to greater severity:
  >70 very atypical 66-70 moderately atypical 61-65 slightly atypical 56-60 borderline range
  ≤ 55 non problematic
Conners' Parent Rating Scale-Revised - Scale K (total CGI) | Before and After 3 months of intervention
  The score of subscale K on the Conners' Parent Rating Scale-Revised reflects a general problem behavior. A high score indicates a hyperactivity problem, often associated with other problem areas.
  The score is a T-score with mean 50 and deviation standard 10 in the general population Minimum score = 35 Maximum score = 100
  Higher scores correspond to greater severity:
  >70 very atypical 66-70 moderately atypical 61-65 slightly atypical 56-60 borderline range
  ≤ 55 non problematic
Conners' Parent Rating Scale-Revised - Scale B (attention problem) | Before and After 3 months of intervention
  Higher scores in the subscale B on the Conners' Parent Rating Scale-Revised are are related to lower learning abilities and difficulties in sustaining prolonged levels of attention.
  The score is a T-score with mean 50 and deviation standard 10 in the general population Minimum score = 35 Maximum score = 100
  Higher scores correspond to greater severity:
  >70 very atypical 66-70 moderately atypical 61-65 slightly atypical 56-60 borderline range
  ≤ 55 non problematic
Conners' Parent Rating Scale-Revised - Scale C ( hyperactivity) | Before and After 3 months of intervention
  Higher scores in the subscale C on the Conners' Parent Rating Scale-Revised are indicative of higher levels of restlessness and impulsivity.
  The score is a T-score with mean 50 and deviation standard 10 in the general population Minimum score = 35 Maximum score = 100
  Higher scores correspond to greater severity:
  >70 very atypical 66-70 moderately atypical 61-65 slightly atypical 56-60 borderline range
  ≤ 55 non problematic
Amyotrophic Lateral Sclerosis Functional Rating Scale - revised (ALSFRS-r) | Before and After 3 months of intervention
  Functional assessment of disease state. maximum score 4 - minimum score 0; for 12 items. indicates normal condition - 0 corresponds to a degree of major severity. The total score can range from a minimum of 0 to a maximum of 48; a score <29 indicates rapid disease progression.
Gastrointestinal Symptom Rating Scale (GSRS) | Before and After 3 months of intervention
  Represents the main symptoms complained about by the patients. maximum score "Unbearable disturbances" - minimum score "No disturbance"; for 15 items.
  The scores follow these directions:
  No disturbance Mild disturbances Bearable disturbances Moderate disturbances Somewhat severe disturbances Severe disturbances Unbearable disturbances
Forced Expiratory Volume - 1st second (FEV1) | Before and After 3 months of intervention
  Expired Volume measured after 1 second during pneumotachography exam
Forced Vital capacity (FVC) | Before and After 3 months of intervention
  Inspired maximal volume during pneumotachography exam
Asthma control test score | Before and After 3 months of intervention
  Test containing items related to cough and breathlessness, validated in asthmatic subjects
  Test contains five items scored on a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled)

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Scientific Institute IRCCS Eugenio Medea, Bosisio Parini, LC
  - Alessia Fumagalli, Casatenovo, LC
  - IBBA-CNR, Milan
  - Centro Clinico NEMO - Fondazione Serena Onlus, Milano, Milan

REFERENCES:
- [Derived] Trezzi S, Scaccabarozzi G, Nossa R, Piazza C, Bianchi AR, Rosi E, Tizzoni F, Mauri M, Camillo L, Baragetti A, Molteni M, Campanella V, Mauro L, Cremonesi P, Severgnini M, Monroy MM, Castiglioni B, Sparvoli F, Pisano S, Pozzi M, Crippa A, Nobile M. Behavioural, cognitive, and neurophysiological effects of a synbiotic supplementation enriched with pigmented corn extract or cornstarch in drug-naive children with attention-deficit hyperactivity disorder: A randomised, double-blind, comparison-controlled clinical trial. Clin Nutr ESPEN. 2025 Feb;65:408-417. doi: 10.1016/j.clnesp.2024.12.016. Epub 2024 Dec 20. PMID 39710171